CLINICAL TRIAL: NCT02320656
Title: Predictive Clinical and Biological Parameters in Acute Leukemia, Myelodysplastic Syndromes and Myeloproliferative Disorders-HEMATO-BIO-IPC-2013-015
Acronym: HEMATO-BIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEMATO-BIO-IPC-2013-015
Record Dates: First submitted 2014-12-05; First posted 2014-12-19 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute leukemia/myelodysplastic or myeloproliferative disease (Experimental)
  Interventions: Other: Blood sampling; Other: Bone marrow aspirate; Other: Skin biopsy; Other: Buccal swab

INTERVENTIONS:
Other: Blood sampling — Longitudinal (3 stages of the disease)
Other: Bone marrow aspirate — Longitudinal (3 stages of the disease)
Other: Skin biopsy — Single biopsy (optional)
Other: Buccal swab — Single sampling.

SUMMARY:
HEMATO-BIO-IPC-2013-015 is a monocenter prospective longitudinal study. Our aim is to define predictive clinical and biological factors in acute leukemia, myelodysplastic syndromes and myeloproliferative disorders by using genomics, genetics and epigenetics, in vitro and in vivo drug sensitivity studies,and translational immonulogy and immunomonitoring studies.

HEMATO-BIO primary outcome measure is to identify molecular, genomic and epigenetic, pharmacologic and immunophenotypic alteration in acute leukemia, myelodysplastic syndromes and myeloproliferative disorders by collecting, at diagnosis and/or complete remission and/or relapse:

* tumor samples: marrow aspiration, blood sampling.
* non-tumor samples: skin biopsy, buccal swab . from 650 patients treated at our cancer center.

ELIGIBILITY:
Inclusion Criteria:

* acute leukemia, myelodysplastic syndrome or myeloproliferative disease
* age > 18
* affiliated to the French Social Security Systm
* signed informed consent

Exclusion Criteria:

* emergency
* patients deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Acute leukemia/ Myeloproliferative/ myelodysplastic syndrome cells profiling (molecular analysis, epigenetic profile, drug sensitivity profile,immunophenotyping) | up to 8 years

SECONDARY OUTCOMES:
Correlation between molecular alteration and clinical characteristics(diagnosis,cytogenetics,overall survival, progression free survival) | up to 8 years
Compare cancer and non-tumor cells genome | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD,PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- [Derived] Grenier JMP, Testut C, Bal M, Bardin F, De Grandis M, Gelsi-Boyer V, Vernerey J, Delahaye M, Granjeaud S, Zemmour C, Spinella JF, Chavakis T, Mancini SJC, Boher JM, Hebert J, Sauvageau G, Vey N, Schwaller J, Hospital MA, Fauriat C, Aurrand-Lions M. Genetic deletion of JAM-C in preleukemic cells rewires leukemic stem cell gene expression program in AML. Blood Adv. 2024 Sep 10;8(17):4662-4678. doi: 10.1182/bloodadvances.2023011747. PMID 38954834
- [Derived] Chretien AS, Devillier R, Granjeaud S, Cordier C, Demerle C, Salem N, Wlosik J, Orlanducci F, Gorvel L, Fattori S, Hospital MA, Pakradouni J, Gregori E, Paul M, Rochigneux P, Pagliardini T, Morey M, Fauriat C, Dulphy N, Toubert A, Luche H, Malissen M, Blaise D, Nunes JA, Vey N, Olive D. High-dimensional mass cytometry analysis of NK cell alterations in AML identifies a subgroup with adverse clinical outcome. Proc Natl Acad Sci U S A. 2021 Jun 1;118(22):e2020459118. doi: 10.1073/pnas.2020459118. PMID 34050021